CLINICAL TRIAL: NCT05260710
Title: Evaluation of the Impact of Telemedicine Use on Clinical Care Indicators in Pediatric Intensive Care Units: Cluster Randomized Controlled Trial
Brief Title: Evaluation of the Impact of Telemedicine in Pediatric Intensive Care Units
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital Moinhos de Vento (Other)
Responsible Party: Principal Investigator, Felipe Cezar Cabral, Digital health coordinator, Hospital Moinhos de Vento
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 5.126.122
Record Dates: First submitted 2022-02-18; First posted 2022-03-02 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Telemedicine; Critical Care; Pediatric; Adolescent; Intensive Care Units, Pediatric
Keywords: Telemedicine; Pediatric Intensive Care Units; Randomized Controlled Clinical Trial; Technology

STUDY DESIGN:
Intervention Model Description: Allocation: Randomized Intervention Model: Parallel Assignment Masking: None (Open Label)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telemedicine intervention (Experimental): Tele-critical care + continuing education activities
  Interventions: Behavioral: Telemedicine Intervention
- Usual Care (No Intervention): Usual Care

INTERVENTIONS:
Behavioral: Telemedicine Intervention — Tele-Critical Care: 1) establishing a diagnosis 2) guiding the therapeutic approach and 3) performing clinical follow-up. Physicians will discuss all patients in the unit, bed by bed, evaluating the specific clinical situation of each hospitalized patient, according to the protocol developed by the study.The proposal is to maintain horizontal care (the patient is monitored from the 1st day of hospitalization until discharge) for all patients in the unit.
  +
  Continuing education activities: video classes and discussions of complex cases.
  Arms: Telemedicine intervention

SUMMARY:
This study will be a cluster randomized controlled trial to assess the impact of telemedicine in Pediatric Intensive Care Units (PICU), through daily tele-rounds with a board certified physician and educational activities, in improving clinical-assistance indicators, as well as reducing the length of stay in the PICU.

DETAILED DESCRIPTION:
This is a parallel cluster randomized controlled trial in pediatric intensive care units in Brazil.

PICUs is the unit of randomization. All patients admitted to the PICUs selected to participate in the project will be included in the study allocated to the control or intervention group as their respective hospitals are randomized.

Intervention group: Tele-rounds are case discussions with remote pediatric intensive care physicians and physicians from other specialties, such as a radiologist, infectious disease specialist, for the debate on conducts based on the best scientific evidence. Additionally, concurrently with the period of application of the intervention, continuing education activities will be made available to all professionals from the teams of the participating centers. Education activities are held monthly and consist of video classes and discussions of complex cases.

Control group: This group will maintain the usual care offered by the participating centers.

ELIGIBILITY:
Inclusion Criteria:

* All children admitted to the pediatric ICU aged ≥29 days and <18 years
* Length of stay of more than 8 hours and, in case of death, with a length of stay of more than 24 hours

Exclusion Criteria:

* Patients with incomplete medical records
* Incomplete data in the institution's database
* Patients whose guardians did not accept to participate in the study and/or who did not sign the informed consent form and the image use term.

Ages: 29 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1760 (Estimated)
Dates: Start 2022-04-01 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Lenght of stay | From PICU admission until the date of PICU discharge or death, whichever comes first, assessed up to 90 days
  Time until discharge from the Pediatric intensive care unit

SECONDARY OUTCOMES:
To measure PICU mortality | From PICU admission until the date of PICU discharge or death, whichever comes first, assessed up to 90 days
  To measure the mortality rate in PICUs
To check the days free from mechanical ventilation | From PICU admission until the date of PICU discharge or death, whichever comes first, assessed up to 90 days
  To check the days free from mechanical ventilation of patients hospitalized in PICUs
To measure the time of use of vasoactive drugs | From PICU admission until the date of PICU discharge or death, whichever comes first, assessed up to 90 days
  To measure the time of use of vasoactive drugs by patients hospitalized in PICUs
To measure the time of use of broad-spectrum antibiotics | From PICU admission until the date of PICU discharge or death, whichever comes first, assessed up to 90 days
  To measure the time of use of broad-spectrum antibiotics in patients hospitalized in PICUs
To measure the time of use of sedation/analgesia | From PICU admission until the date of PICU discharge or death, whichever comes first, assessed up to 90 days
  To measure the time of use of sedation/analgesia in patients hospitalized in PICUs

CONTACTS AND LOCATIONS:
Overall Officials: Felipe C Cabral, Principal Investigator — Hospital Moinhos de Vento

IPD SHARING:
Plan to Share IPD: Yes
With the publication of the main study the IPD will be available to researchers not members of the study.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will become available with the publication of the main study.
Access Criteria: Data will be acessed through an online repository protected with password and for secondary analyses according to pre-specified plans.

REFERENCES:
- [Background] Agência IBGE https://agenciadenoticias.ibge.gov.br/agencia-noticias/2012-agencia-de-notíci as/27614-ibge-divulga-distribuicao-de-utis-respiradores-medicos-e-enfermeiros: Acessado em 14 de novembro de 2020.
- [Background] BRASIL. Ministério da Saúde. Diretrizes Operacionais para o Estabelecimento e o Funcionamento de Comitês de Monitoramento de Dados e de Segurança / Ministério da Saúde, Organização Mundial da Saúde. Brasília : Ministério da Saúde, 2008. 44 p.
- [Background] Campbell MK, Piaggio G, Elbourne DR, Altman DG; CONSORT Group. Consort 2010 statement: extension to cluster randomised trials. BMJ. 2012 Sep 4;345:e5661. doi: 10.1136/bmj.e5661. No abstract available. PMID 22951546
- [Background] Chen J, Sun D, Yang W, Liu M, Zhang S, Peng J, Ren C. Clinical and Economic Outcomes of Telemedicine Programs in the Intensive Care Unit: A Systematic Review and Meta-Analysis. J Intensive Care Med. 2018 Jul;33(7):383-393. doi: 10.1177/0885066617726942. Epub 2017 Aug 22. PMID 28826282
- [Background] DE AZEVEDO, Arimatéia Portela et al. Fatores que interferem no desempenho da utilização de leitos de unidade de terapia intensiva (UTI). Brazilian Journal of Health Review, v. 3, n. 4, p. 7421-7438, 2020.
- [Background] Garingo A, Friedlich P, Chavez T, Tesoriero L, Patil S, Jackson P, Seri I. "Tele-rounding" with a remotely controlled mobile robot in the neonatal intensive care unit. J Telemed Telecare. 2016 Mar;22(2):132-8. doi: 10.1177/1357633X15589478. Epub 2015 Jun 26. PMID 26116855
- [Background] Grundy BL, Crawford P, Jones PK, Kiley ML, Reisman A, Pao YH, Wilkerson EL, Gravenstein JS. Telemedicine in critical care: an experiment in health care delivery. JACEP. 1977 Oct;6(10):439-44. doi: 10.1016/s0361-1124(77)80239-6. PMID 71365
- [Background] MINISTÉRIO DA SAÚDE. Portaria n. 3.432, de 12 de agosto de 1998. Estabelece Critérios de Classificação de Unidade de Terapia Intensiva (UTI). Diário Oficial da União n. 154; Poder Executivo, 13 ago. 1998. Disponível em: <www.medicinaintensiva.com.br/portaria-3432.htm>. Acesso em: 10 jan. 2010.
- [Background] Moher D, Hopewell S, Schulz KF, Montori V, Gotzsche PC, Devereaux PJ, Elbourne D, Egger M, Altman DG; CONSORT. CONSORT 2010 explanation and elaboration: updated guidelines for reporting parallel group randomised trials. Int J Surg. 2012;10(1):28-55. doi: 10.1016/j.ijsu.2011.10.001. Epub 2011 Oct 12. PMID 22036893
- [Background] PATRIDGE, Emily F.; BARDYN, Tania P. Research electronic data capture (REDCap). Journal of the Medical Library Association: JMLA, v. 106, n. 1, p. 142, 2018.
- [Background] PARK, Heesun. SAS Institute, Inc. Cary, North Carolina. Sign, v. 2, n. 4, p. 1.
- [Background] Pfrimmer DM, Roslien JJ. The Tele-ICU: a new dimension in critical care nursing education and practice. J Contin Educ Nurs. 2011 Aug;42(8):342-3. doi: 10.3928/00220124-20110722-03. PMID 21800788
- [Background] Piaggio G, Elbourne DR, Pocock SJ, Evans SJ, Altman DG; CONSORT Group. Reporting of noninferiority and equivalence randomized trials: extension of the CONSORT 2010 statement. JAMA. 2012 Dec 26;308(24):2594-604. doi: 10.1001/jama.2012.87802. PMID 23268518
- [Background] Jacovas VC, Chagas MEV, Constant HMRM, Alves SS, Krauzer JRM, Guerra LR, de Almeida Pires A, Gomes da Cunha L, Matte MCC, de Campos Moreira T, Cabral FC. Telemedicine in Pediatric Intensive Care Units: Perspectives From a Brazilian Experience. Curr Pediatr Rep. 2021;9(3):65-71. doi: 10.1007/s40124-021-00242-z. Epub 2021 Jul 12. PMID 34277142
- [Derived] de Oliveira Laguna Silva G, Konig Klever E, Castro da Rocha J, da Silva MMD, da Rosa de Amorim J, Cristina Jacovas V, Marina Simionato B, Gomes da Cunha L, Zaupa APB, Mafalda Krauzer JR, de Almeida Pires A, Cezar Cabral F, de Campos Moreira T, Rodrigues Moleda Constant HM. Evaluation of the use of telemedicine in pediatric intensive care units: a cluster-randomized trial. Postgrad Med. 2024 Aug;136(6):633-640. doi: 10.1080/00325481.2024.2388023. Epub 2024 Aug 5. PMID 39093639
- [Derived] Silva MMDD, Klever EK, Rocha JCD, Silva GOL, Amorim JDR, Dode AD, Simionato BM, Cunha LGD, Zaupa APB, Krauzer JRM, Pires AA, Cabral FC, Moreira TC, Constant HMRM. Impact of Telemedicine use on clinical care indicators of pediatric intensive care units: protocol for a cluster randomized clinical trial. Crit Care Sci. 2023 Dec 22;35(3):266-272. doi: 10.5935/2965-2774.20230223-en. eCollection 2023. PMID 38133156